CLINICAL TRIAL: NCT02723877
Title: An Open Label, Non Randomized, Multicenter Phase 1/2b Study Investigating Safety and Efficacy of PQR309 and Eribulin Combination in Patients With Locally Advanced or Metastatic HER2 Negative and Triple-Negative Breast Cancer
Brief Title: PQR309 and Eribulin in Metastatic HER2 Negative and Triple-negative Breast Cancer (PIQHASSO)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PIQUR Therapeutics AG (Industry)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Hospital Universitari Vall d'Hebron Research Institute (Other); Institut Català d'Oncologia (Other); Churchill Hospital (Other); Barts Cancer Institute (Other); Fundación Instituto Valenciano de Oncología (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQR309-007
Record Dates: First submitted 2015-12-21; First posted 2016-03-31 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Breast Cancer
Keywords: TNBC
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eribulin and PQR309 (Experimental): PQR309 in combination with standard approved dose of eribulin mesylate 1.4 mg/m2 intravenous (iv) on days 1 and 8 in a period of 21 days per cycle will be investigated. . PQR309 will be administered maximum 15 minutes after eribulin iv dosing.
  Interventions: Drug: PQR309; Drug: Eribulin

INTERVENTIONS:
Drug: PQR309 — Dual phosphatidylinositol 3-kinase phosphoinositide 3-kinase/ mammalian target of rapamycin Inhibitor (= PI3K/mTOR Inhibitor)
Drug: Eribulin — non.taxane microtubule dynamics inhibitor
  Other Names: eribulin mesylate; Halaven®

SUMMARY:
This study is an open-label,non randomized, multi-center, phase 1/2b (dose escalation followed by expansion part) study evaluating clinical safety, efficacy and pharmacokinetics of PQR309 in combination with standard dose of eribulin in patients with locally advanced or metastatic HER2-negative (escalation part) and Triple Negative Breast Cancer (expansion part).

DETAILED DESCRIPTION:
* The primary objective of the escalation part is to assess the maximum tolerated dose (MTD) of PQR309 combined with the standard eribulin dose in patients with HER2 negative breast cancer following a "modified" 3 by 3 design.
* For the expansion part the objective is to evaluate efficacy of PQR309 in combination with eribulin in patients with Triple Negative Breast Cancer
* Once the MTD of continuous daily PQR309 dosing has been established, intermittent schedules of PQR309 ("2 days on/ 5 days off" or "Monday / Thursday") will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed diagnosis of breast cancer. Radiological evidence of inoperable locally advanced or metastatic breast cancer.
* HER2 negative breast cancer (based on the most recent analyzed biopsy) defined as a negative in situ hybridization test or an immunohistochemistry status of 0, 1+ or 2+.
* Received at least 2 and no more than 5 prio chemotherapeutic regimens in locally advanced and/or metastatic setting.
* Prior therapy has to include an anthracycline and a taxane in any combination or order.
* For Expansion part:

Triple-negative breast cancer defined as a negative in situ hybridization test or an immunohistochemistry (IHC) status of 0,1+ or 2+ER abnd PR status <10% by local laboratory testing.

Exclusion Criteria:

* Previous systemic treatment with PI3K,mTOR or AKT inhibitors (allowed in the escalation part).
* Previous treatment with eribulin (allowed in the escalation part). Known hypersensitivity to any of the excipients of PQR309 or eribulin.Concurrent treatment with other approved or investigational antineoplastic agent.
* Symptomatic Central Nervous System metastases. The patient must have completed any prior local treatment for CNS metastases > 28 days prior to first dose of the study drug (including radiotherapy and/or surgery).
* Clinically manifested diabetes mellitus(treated and/or clinical signs with fasting glucose >125mg/dl or HbA1c>7%), or documented steroid induced diabetes mellitus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment related Adverse Events and Serious Adverse Events as assessed by NCI CTCAEV4.03 | Up to 6 months
  Continous dosing and intermittent schedules of PQR309
RECIST the Response criteria for solid tumors will be used to identify clinical benefit rate (CBR) including complete Response (CR), partial Response (PR) and stable disease (SD) | Up to 15 months
  Continous dosing and intermittent schedules of PQR309

SECONDARY OUTCOMES:
Number of patients with Adverse Events and Serious Adverse Events and number of anormal laboratory values that constitute an Adverse Events on their own | Up to 12 months
  Continous dosing and intermittent schedules of PQR309
Number and percent of patients having each ECOG (Eastern Oncology Cooperative Group) performance status level will be presented for baseline and each post-baseline measurement. | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Assessment of PQR309 and Eribulin blood concentration | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Physical examination, Body weight in kg | up to 12 months
  Continous dosing and intermittent schedules
Physical examination, ECG | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Vital signs like heart rate | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Vital signs like blood pressure | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Vital signs like body temperature | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Objective Response Rate (ORR), is defined as the best overall response (confirmed CR or PR) recorded for each patient since baseline. | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Time to Response (TTR) is defined, for patients with tumor response, as the time from the date of study entry to the first documentation of response (complete or partial) | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Duration of response (DOR) is defined, for the patients with tumor response, as the time from the date of the first confirmed response to disease progression. | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Progression- free survival (PFS) is defined as the time from study entry to progression or death due to any cause | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Time to treatment failure (TTF) is defined as the time from study entry to any treatment failure including disease progression or discontinuation of treatment | up to 12 months
  Continous dosing and intermittent schedules of PQR309
1-year survival, defined as the time from study entry to death as a result of any cause at 1-year cut-off date | up to 12 months
  Continous dosing and intermittent schedules of PQR309
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: tmax | On Cycle 1 Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion and on Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose
  Intermittent schedule B: "Monday/ Thursday"
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: cmax | On Cycle 1 Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion and on Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose
  Intermittent schedule B: "Monday/ Thursday"
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: AUC0-24 | On Cycle 1 Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion and on Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose
  Intermittent schedule B: "Monday/ Thursday"
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: AUC0-∞ | On Cycle 1 Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion and on Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose
  Intermittent schedule B: "Monday/ Thursday"
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: RAC(Racemate) | On Cycle 1 Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion and on Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose
  Intermittent schedule B: "Monday/ Thursday"
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: cmax | PK is being assessed during Cycle 1 on Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion. On Cycle 1 Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose.
  Intermittent schedule A: 2 days on/5 days off
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: tmax | PK is being assessed during Cycle 1 on Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion. On Cycle 1 Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose.
  Intermittent schedule A: 2 days on/5 days off
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: AUC0-24 | PK is being assessed during Cycle 1 on Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion. On Cycle 1 Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose.
  Intermittent schedule A: 2 days on/5 days off
PK parameters of PQR309 and eribulin will include: AUC0-∞ | PK is being assessed during Cycle 1 on Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion. On Cycle 1 Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose.
  Intermittent schedule A: 2 days on/5 days off
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: RAC | PK is being assessed during Cycle 1 on Day 8: pre-dose, end of eribulin infusion, 2h and 6h post end of eribulin infusion. On Cycle 1 Day 15: pre-dose and one sample between 1 and 3 hours post PQR309 dose.
  Intermittent schedule A: 2 days on/5 days off
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: cmax | It will be measured pre-dose and at the end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end and at end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end of eribulin during Cycle 1 on day 1 and 8 and beyond cycle 1 on day 1
  Continous Dosing
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: AUC0-24 | It will be measured pre-dose and at the end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end and at end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end of eribulin during Cycle 1 on day 1 and 8 and beyond cycle 1 on day 1
  Continous Dosing
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: AUC0-∞ | It will be measured pre-dose and at the end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end and at end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end of eribulin during Cycle 1 day on 1 and 8 and beyond cycle 1 on day 1
  Continous Dosing
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: t1/2 | It will be measured pre-dose and at the end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end and at end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end of eribulin during Cycle 1 on day 1 and 8 and beyond cycle 1 on day 1
  Continous Dosing
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: tmax | It will be measured pre-dose and at the end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end and at end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end of eribulin during Cycle 1 on day 1 and 8 and beyond cycle 1 on day 1
  Continous Dosing
Pharmacokinetic (PK) parameters of PQR309 and eribulin will include: RAC (Racemate) | It will be measured pre-dose and at the end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end and at end of eribulin infusion and 0.5h, 1h, 2h, 4h, and 8h post end of eribulin during Cycle 1 on day 1 and 8 and beyond cycle 1 on day 1
  Continous Dosing
Changes in glucose levels | 12 months
  Continous dosing and intermittent schedules of PQR309
Changes in Insulin levels | 12 months
  Continous dosing and intermittent schedules of PQR309
Changes of Routine laboratory -Haematology | 12 months
  Continous dosing and intermittent schedules of PQR309
Changes of Routine laboratory -blood chemistry | 12 months
  Continous dosing and intermittent schedules of PQR309
Changes of Routine laboratory -urinanalysis | 12 months
  Continous dosing and intermittent schedules of PQR309

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortes, PD Dr. med, Study Director — Hospital Universitario Ramon y Cajal
Locations (5):
- Spain (3):
  - Hospital Universitarsi Vall d'Hebron, Barcelona, Catalan
  - Insitut Català d´Oncologia, Barcelona
  - Fundación Instituto Valenciano de Oncología, Valencia
- United Kingdom (2):
  - Barts Cancer Institute, London
  - Churchill hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided